CLINICAL TRIAL: NCT04637503
Title: Multi-center Phase I/II Clinical Trial of 4SCAR-T Therapy Targeting GD2, PSMA and CD276 for Treating Neuroblastoma
Brief Title: 4SCAR-T Therapy Targeting GD2, PSMA and CD276 for Treating Neuroblastoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: Shenzhen Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-20010
Record Dates: First submitted 2020-10-16; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Neuroblastoma
Keywords: CART; chimeric antigen receptor; adoptive T cell transfer; GD2, PSMA, CD276, B7-H3
MeSH Terms: conditions — Neuroblastoma; Gaucher Disease | interventions — ganglioside, GD2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- effectiveness of CAR-T cells targeting GD2, PSMA and CD276 (Experimental): Gene-modified T cells are designed to kill tumor cells through specific recognition of GD2, PSMA and CD276. This study will evaluate the side effects and effective doses of GD2, PSMA and CD276 CAR-T cells in treating refractory and recurrent NB
  Interventions: Biological: GD2, PSMA and CD276 CAR-T cells

INTERVENTIONS:
Biological: GD2, PSMA and CD276 CAR-T cells — infusion, for 1x10^6~1x10^7 cells/kg via IV

SUMMARY:
The purpose of this clinical trial is to assess the feasibility, safety and efficacy of multiple 4SCAR-T cell therapy which targets GD2, PSMA and CD276 surface antigens in patients with relapsed and refractory neuroblastoma (NB). Another goal of the study is to understand the function of the multi-CAR-T cells and their persistency in the patients.

DETAILED DESCRIPTION:
Neuroblastoma is one of the most aggressive childhood tumors arising from neural crest cells. Nearly 50% of patients with high risk disease have poor long-term survival even after multimodal treatments. Novel immunotherapy targeting tumor-specific antigens has been developed to meet the desperate need.

Disialoganglioside (GD2) is a well-studied tumor associated antigen which is expressed uniformly in NB but restrictedly in normal tissue. Over the past few years, CAR-T therapy against GD2 in NB has achieved encouraging but modest outcomes. Only a fraction of patients achieved measurable responses. Like for many other solid tumors, CAR-T therapy for NB is not as effective as for hematologic malignancies.

In this study, the investigators use "multiple targeting" approach as the strategy to overcome the challenge in treating NB. Prostate-specific membrane antigen (PSMA) is expressed in normal prostate but is upregulated in prostate tumor. However, PSMA expression is not restricted to prostate cancer. By immunohistochemistry (IHC) staining, the investigators confirmed that PSMA is expressed in a variety of solid tumors, including brain tumor, neuroblastoma and some lymphoma tumor tissues. Therefore, PSMA could potentially serve as a promising target for antigen-specific immunotherapy in patients with NB. In addition, CD276 (B7-H3) is an immune checkpoint molecule highly expressed on many solid tumors including NB. CD276 has been characterized to be involved in tumor evasion and thus its expression is correlated with poor prognosis. These characteristics make CD276 an attractive candidate for immunotherapy. Given the significant variation of tumor antigen expression among patients, the investigators aim to examine GD2, PSMA and CD276 expression in each patient's tumor sections by IHC staining, and combine two or three highly-expressed targets for the 4SCAR-T therapy. This individualized and multi-antigen-targeted approach is a new strategy to overcome the limited clinical outcome in the 4SCAR-T therapy against NB.

The purpose of this clinical study is to assess the feasibility, safety and efficacy of the combinational GD2, PSMA and CD276 4SCAR-T cell therapy against NB. Another goal of the study is to learn more about the function of the multi-4SCAR-T cells and their persistency in the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumors have received standard first-line therapy and been judged to be non-resectable, metastatic, progressive or recurrent.
* The expression status of GD2, PSMA and CD276 antigens of the tumor will be determined for eligibility. Positive expression is defined by GD2, PMSA and CD276 antibody staining results based on immunohistochemistry or flow cytometry analyses.
* Body weight greater than or equal to 10 kg.
* Age: ≥1 year and ≤ 65 years of age at the time of enrollment.
* Life expectancy: at least 8 weeks.
* Prior Therapy:

  1. There is no limit to the number of prior treatment regimens. Any grade 3 or 4 non-hematologic toxicity of any previous therapy must have resolved to grade 2 or less.
  2. Participant must not have received hematopoietic growth factors for at least 1 week prior to mononuclear cells collection.
  3. At least 7 days must have elapsed since the completion of therapy with a biologic agent, targeted agent, tyrosine kinase inhibitor or a metronomic non-myelosuppressive regimen.
  4. At least 4 weeks must have elapsed since prior therapy that included a monoclonal antibody.
  5. At least 1 week since any radiation therapy at the time of study entry.
* Karnofsky/jansky score of 60% or greater.
* Cardiac function: Left ventricular ejection fraction greater than or equal to 40/55 percent.
* Pulse Ox greater than or equal to 90% on room air.
* Liver function: defined as alanine transaminase (ALT) <3x upper limit of normal (ULN), aspartate aminotransferase (AST) <3x ULN; serum bilirubin and alkaline phosphatase <2x ULN.
* Renal function: Patients must have serum creatinine less than 3 times upper limit of normal.
* Marrow function: White blood cell count ≥1000/ul, Absolute neutrophil count ≥500/ul, Absolute lymphocyte count ≥500/ul, Platelet count ≥25,000/ul (not achieved by transfusion).
* Patients with known bone marrow metastatic disease will be eligible for study as long as they meet hematologic function criteria, and the marrow disease not evaluable for hematologic toxicity.
* For all patients enrolled in this study, their parents or legal guardians must sign an informed consent and assent.

Exclusion Criteria:

* Existing severe illness (e.g. significant cardiac, pulmonary, hepatic diseases, etc.) or major organ dysfunction, with the exception of grade 3 hematologic toxicity.
* Untreated central nervous system (CNS) metastasis: Patients with previous CNS tumor involvement that has been treated and is stable for at least 6 weeks following completion of therapy are eligible.
* Previous treatment with other genetically engineered GD2, PSMA and CD276 CART cells.
* Active HIV, Hepatitis B virus (HBV), Hepatitis C virus (HCV) infection or uncontrolled infection.
* Patients who require systemic corticosteroid or other immunosuppressive therapy.
* Evidence of tumor potentially causing airway obstruction.
* Inability to comply with protocol requirements.
* Insufficient CART cells availability.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-18 (Estimated); Primary Completion 2020-11-19 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | 3 year
  Determine the toxicity profile the GD2, PSMA and CD276 4SCAR-T cells with Common Toxicity Criteria for Adverse Effects version 4.0

SECONDARY OUTCOMES:
Anti-tumor effects | 3 year
  Complete response/remission (CR), Very good partial response/remission (VGPR) will be assessed by the image scan
The expansion of CAR-T cells | 3 year
  The investigators will monitor the expansion of GD2, PSMA and CD276 CAR-T cells in the peripheral blood of patients and the correlation with antitumor effects.
The anti-tumor activity after CAR-T infusions | 1 year
  The anti-tumor activity of lymphocytes will be assessed
The cytokine secretion profile after CAR-T infusions | 1 year
  The cytokine secretion profile of lymphocytes will be assessed.
Survival time of the patients | 3 year
  The overall survival time of the patients treated with CAR-T cells

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Guangdong Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Shenzhen Geno-Immune Medical Institute, Shenzhen, Guangzhou
  - Shandong Cancer Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No